CLINICAL TRIAL: NCT00966277
Title: Randomized Clinical Trial of Dalteparin for Primary Venous Thromboembolism (VTE) Prophylaxis in Pancreatic Cancer Patients Undergoing Chemotherapy Treatment.
Brief Title: Dalteparin for Primary Venous Thromboembolism (VTE) Prophylaxis in Pancreatic Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0487; NCI-2011-01773 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Pancreatic Cancer; Venous Thromboembolism
Keywords: Pancreas; Primary venous thromboembolism; VTE; Chemotherapy; Deep venous thrombosis; Pulmonary embolism; Dalteparin; Fragmin; Thromboprophylaxis
MeSH Terms: conditions — Pancreatic Neoplasms; Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Dalteparin (Experimental): Dalteparin 5000 units subcutaneous, by injection under the skin, daily for 16 weeks.
  Interventions: Drug: Dalteparin
- Group 2: Control (No Intervention): No study drug.

INTERVENTIONS:
Drug: Dalteparin — 5000 units subcutaneous, by injection under the skin, daily for 16 weeks
  Other Names: Fragmin
  Arms: Group 1: Dalteparin

SUMMARY:
The goal of this clinical research study is to learn if dalteparin can lower the risk of VTE occurring in the legs and lungs. This will be tested in patients with pancreatic cancer who are going to receive chemotherapy. Some patients will receive dalteparin and some will receive no study drug.

The safety of dalteparin will also be studied.

DETAILED DESCRIPTION:
Study Drug:

Dalteparin is designed to thin the blood and block blood from clotting. This may lower the risk of VTE.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) into 1 of 2 groups. There is an equal chance of being assigned to either group.

Group 1 will receive dalteparin.

Group 2 will not receive a study drug.

During this study, all study participants will be routinely checked for VTE by ultrasounds and CT scans.

You may also receive standard therapies for preventing VTE. This may include blood-thinning drugs while you are in the hospital, getting up and moving around at least 5 times per day, and/or wearing special stockings or boot-like devices designed to put pressure on the feet.

Genetic Research Testing:

Before starting your therapy (at baseline), blood (about 1 teaspoon) will be drawn and stored for genetic testing. Researchers want to use DNA (the genetic material in cells) to look for markers that may be related to having a high risk for developing blood clots. The samples will be processed and stored at MD Anderson. Once this study ends, the DNA will be tested further in Dr. Futreal's laboratory and/or may be shipped outside to Illumina Sequencing Services (San Diego, CA) for genetic research. The samples will be deidentified before shipping.

Before your samples are sent to the outside laboratory for banking, your name and any personal identifying information will be coded to protect your privacy. The outside researchers will not have access to the codes that link the samples to your identity.

Study Drug Administration:

If you are in Group 1, you will receive dalteparin by injection under your skin, once a day for 16 weeks. You and/or your caregiver will be taught how to perform injections.

Study Visits:

At every study visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature and breathing rate).
* Your medical history will be recorded.

About every 2 weeks after chemotherapy starts until Week 16, blood (about 2 teaspoons) will be drawn for routine tests. This test may be repeated more often if the doctor decides it is needed.

Before each new cycle of chemotherapy during Weeks 1-16, blood (about 2 teaspoons) will be drawn for routine tests to check the function of your liver and kidneys.

At Weeks 8 and 16 (+/- 7 days), the following procedures will be performed:

* You will have an ultrasound of your legs to check for blood clots.
* If the doctor decides it is needed, you will have CT scans to check the status of the cancer. Researchers will also check your chest CT scans to look for blood clots in the lungs.

Length of Study Participation:

You may remain on study for up to 16 weeks. You will be taken off study early if blood clots occur or you experience intolerable side effects.

Follow-Up Phone Calls:

This study has a 3-year follow-up period. In Year 1, you will receive a follow-up phone call from the study staff in the first month and then at Months 3, 6, 9, and 12. In Years 2 and 3, you will be called every 6 months.

The study staff will ask about your overall health. In the first phone call, you will also be asked about any side effects that may have occurred.

This is an investigational study. Dalteparin is commercially available and FDA approved for use in preventing VTE that may occur for other reasons. Those reasons include abdominal surgery; surgery for a hip fracture, hip replacement, or knee replacement; and illnesses causing patients to be unable to move around.

Dalteparin is also commercially available and FDA approved to treat VTE in cancer patients. However, it is investigational to use dalteparin to prevent VTE in cancer patients receiving chemotherapy.

Up to 87 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnosis of advanced stage (unresectable or metastatic) adenocarinoma of the pancreas. Patients with borderline resectable will also be eligible if they are starting chemotherapy and/or chemo/radiation therapy (RT) prior to attempting resection.
2. Patients must be planning to initiate systemic chemotherapy within 2 weeks. Chemotherapy that is being given concurrently with radiation is allowed.
3. Age >/= 18 years old
4. Adequate renal function defined as a calculated creatinine clearance of > 50 mL/min (as reported by the MDACC laboratory using MDRD method or using Cockroft and Gault formula).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
6. Negative urine or serum pregnancy test in women with childbearing potential, within one week prior to initiation of treatment.
7. Patients must sign an Informed Consent.
8. Patient must agree to transfusion of blood products, when indicated.
9. Ability to administer subcutaneous injections of the study drug by the patient and/or care giver.

Exclusion Criteria:

1. Patients with evidence of venous thrombosis on the initial lower extremity screening ultrasound or incidental VTE of other sites (e.g. PE, Abdominal/pelvic vein thrombosis, etc.).
2. Patients already taking prophylactic or full dose anticoagulation (eg. heparin, low-molecular weight heparin, fondaparinux, or coumadin).
3. Patients with currently active bleeding.
4. The presence of a condition with a high risk for bleeding, including but not limited to active peptic ulcer, recent neurosurgery, or cirrhosis with esophageal varices.
5. Patients with known brain metastases.
6. Patients with a known bleeding diathesis.
7. Patients with a platelet count < 50,000.
8. Patients with known hypersensitivity to dalteparin.
9. Patients who regularly use medications known to increase the risk of bleeding such as >/= 325 mg of aspirin daily, or daily clopidogrel, or daily non-steroidal antiinflammatory medications (eg., ibuprofen, naproxen).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kahale LA, Matar CF, Hakoum MB, Tsolakian IG, Yosuico VE, Terrenato I, Sperati F, Barba M, Schunemann H, Akl EA. Anticoagulation for the initial treatment of venous thromboembolism in people with cancer. Cochrane Database Syst Rev. 2021 Dec 8;12(12):CD006649. doi: 10.1002/14651858.CD006649.pub8. PMID 34878173
- [Derived] Kahale LA, Matar CF, Tsolakian I, Hakoum MB, Barba M, Yosuico VE, Terrenato I, Sperati F, Schunemann H, Akl EA. Oral anticoagulation in people with cancer who have no therapeutic or prophylactic indication for anticoagulation. Cochrane Database Syst Rev. 2021 Oct 8;10(10):CD006466. doi: 10.1002/14651858.CD006466.pub7. PMID 34622445
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: April 06, 2010 to August 23, 2012. All recruitment done at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 87 participants enrolled on the study, only 75 were randomized. Twelve enrolling participants were screen failures or withdrew before randomization thus were excluded before assignments to groups.
Groups:
- Group 2: Control: No Dalteparin study drug (primary prophylaxis).
Period: Overall Study
Arm/Group | Group 1: Dalteparin | Group 2: Control
Started | 38 | 37
Completed | 34 (Four participants did not receive study treatment, see 'Reasons Not Completed.') | 33 (Four participants did not receive study treatment, see 'Reasons Not Completed.')
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Ineligible | 1 | 3
Not completed — Treatment Plan Changed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Control: No Dalteparin study drug.
- Total: Total of all reporting groups
Arm/Group | Group 1: Dalteparin | Group 2: Control | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Continuous [Mean (Full Range); unit: years] | 59 [36 to 75] | 64 [38 to 77] | 61.5 [36 to 77]
Age, Customized [Number; unit: years]
  <60 | 21 | 10 | 31
  >=60 | 17 | 27 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 20 | 21 | 41
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 2 | 5
  Causacian | 31 | 31 | 62
  Hispanic | 2 | 3 | 5
  Other | 1 | 0 | 1
  Unknown or Unreported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Venous Thromboembolic Events (VTE)
Description: Venous thromboembolism (VTE) defined by both symptomatic and asymptomatic VTE which includes deep venous thrombosis (DVT) and pulmonary embolism (PE) through clinical assessments and radiologic studies. All patients undergo bilateral lower extremity ultrasound every 2 months while on study (total of 3 exams including pre-randomization). VTE requires imaging documentation to evaluate use of prophylactic anticoagulation in reducing the occurrence of VTE in a patient population with a known high risk of VTE.
Time Frame: 16 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Group 1: Dalteparin | Group 2: Control
Number analyzed (Participants) | 38 | 37
participants | 2 | 9

ADVERSE EVENTS:
Time Frame: Follow-up/observation for all adverse events will be through Day 28 following the last dose of study drug or until resolution of any toxicity related to the study drug at the end of treatment.
Arm/Group | Group 1: Dalteparin | Group 2: Control
Serious Adverse Events (participants affected / at risk) | 34/34 | 33/33
Other Adverse Events (participants affected / at risk) | 34/34 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Dalteparin (N=34) | Group 2: Control (N=33)
Vomiting (Gastrointestinal disorders) | 15 | 7
Constipation (Gastrointestinal disorders) | 16 | 9
Abdominal pain (Gastrointestinal disorders) | 12 | 7
Nausea (Gastrointestinal disorders) | 20 | 15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Dalteparin (N=34) | Group 2: Control (N=33)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Anxiety (Psychiatric disorders) | 4 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Bruising/minor bleeding (Injury, poisoning and procedural complications) | 8 | 2 — Grade 1
Depression (Psychiatric disorders) | 1 | 8
Dermatology/Skin (Other) (Skin and subcutaneous tissue disorders) | 2 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Bruising/Bleeding (Injury, poisoning and procedural complications) | 0 | 1 — Grade 2/3
Insomnia (Psychiatric disorders) | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 10
Ocular/Visual (Other) (Eye disorders) | 2 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Pulmonary (Other) (Respiratory, thoracic and mediastinal disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes